CLINICAL TRIAL: NCT02856113
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Alogliptin Compared With Placebo in Pediatric Subjects With Type 2 Diabetes Mellitus
Brief Title: Phase 3 Alogliptin Pediatric Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYR-322_309; U1111-1174-1923 (Registry Identifier: WHO); 2015-000208-25 (EudraCT Number); 173300410A0019 (Registry Identifier: NREC); MOH_2017-12-26_000698 (Other: CRS)
Record Dates: First submitted 2016-08-02; First posted 2016-08-04 (Estimated); Results first posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — alogliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Alogliptin matching-placebo tablets, orally, once daily (QD) for 52 weeks and background antidiabetic therapy (metformin and/or insulin), if applicable, maintained at the same dose throughout the first 26 weeks of the treatment period.
  Interventions: Drug: Placebo
- Alogliptin 25 mg (Experimental): Alogliptin 25 mg tablets, orally, QD for 52 weeks and background antidiabetic therapy (metformin and/or insulin), if applicable, maintained at the same dose throughout the first 26 weeks of the treatment period.
  Interventions: Drug: Alogliptin Benzoate

INTERVENTIONS:
Drug: Alogliptin Benzoate — Alogliptin benzoate tablets.
  Other Names: SYR-322; Nesina; Vipidia
  Arms: Alogliptin 25 mg
Drug: Placebo — Alogliptin placebo-matching tablets.
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to evaluate the efficacy of alogliptin 25 milligram (mg) once daily compared to placebo when administered as monotherapy, or when added onto a background of metformin alone, insulin alone, or a combination of metformin and insulin, as measured by the glycosylated hemoglobin (HbA1c) change from Baseline at Week 26 in pediatric participants with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
The drug being tested in this study is called alogliptin. Alogliptin is being tested to treat children 10 to 17 years of age who have T2DM and are experiencing inadequate glycemic control. This study will look at HbA1c fluctuations in children who take alogliptin in addition to their background antidiabetic therapy.

The study will enroll approximately 150 participants. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups-which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* Alogliptin 25 mg
* Placebo (dummy inactive pill) - this is a tablet that looks like the tablet containing alogliptin 25 mg but has no active ingredient (that is, has no alogliptin).

All participants will be asked to take one tablet at the same time each day throughout the study in addition to their current background antidiabetic therapy (metformin and/or insulin) if applicable.

This multi-center trial will be conducted worldwide. The overall time to participate in this study is approximately 56 weeks. Participants will make multiple visits to the clinic, and will be contacted by telephone 2 weeks after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Has a confirmed diagnosis of T2DM using American Diabetes Association (ADA) and World Health Organization (WHO) criteria (laboratory determinations of fasting plasma glucose [FPG] greater than or equal to [>=] 126 mg/dL, random glucose >=200 mg/dL [>=11.10 mmol/L], HbA1c >=6.5 percent (%), or 2-hour oral glucose tolerance test [OGTT] glucose >=200 mg/dL), documented in the participants' medical record.
2. The participant and/or his/her legal representative (that is, parents or legal guardians) are able and willing to monitor their own blood glucose concentrations with a home glucose monitor and complete participant diaries.

Exclusion Criteria:

1. Has a history of hypersensitivity or allergy to alogliptin, other dipeptidyl peptidase-4 (DPP-4) inhibitors, metformin, insulin or related compounds.
2. Has a confirmed diagnosis of type 1 diabetes mellitus or maturity-onset diabetes of the young (MODY).
3. Has a hemoglobin level <11.0 gram per deciliter (g/dL) (<110 gram per liter [g/L]) for males and <10.0 g/dL (<100 g/L) for females.
4. Has a history of any hemoglobinopathy that may affect determination of HbA1c levels.
5. Has a history of bariatric surgery.
6. Has a history of proliferative diabetic retinopathy within the 6 months prior to Screening.
7. Has had more than 1 episode of diabetic ketoacidosis (DKA) at any time after diagnosis of T2DM.
8. Has a history of more than 1 episode of pancreatitis.
9. Has serum creatinine >=1.5 mg/dL for male participants or >=1.4 mg/dL for female participants, or creatinine clearance <60 milliliter per minute (mL/min) based on calculation by central lab using the Schwartz formula for estimated glomerular filtration rate (eGFR) at screening Visit.
10. Has a documented history of infection with human immunodeficiency virus or chronic active viral hepatitis.
11. The participant and/or his/her legal representative (that is, parents or legal guardians) is unable to understand verbal or written English, or any other language for which a certified translation of the approved informed consent/assent is available.

Additional Criteria That Must be Met Prior to Randomization:

For participants who have had the diagnosis of T2DM for less than 1 year and/or who are taking insulin at Screening, additional criteria will need to be met prior to randomization:

1. Must have an HbA1c level of >=6.5% to <11.0% if the participant is treatment naïve or on metformin alone or >=7.0% to <11.0% if the participant is on insulin alone or in combination with metformin.
2. The participant must not have received any investigational compound within 30 days or 5 half-lives, whichever is longer, prior to randomization.
3. Must not have received an antidiabetic agent other than metformin or insulin within the 12 weeks prior to randomization.
4. Must not have received oral or parenteral steroids for more than 3 weeks (cumulatively) within the 6 months prior to randomization or have received a course of oral or parenteral steroids within the 2 months prior to randomization.
5. Has a systolic blood pressure <160 millimeter of mercury (mmHg) and a diastolic pressure <100 mm Hg. (Antihypertensive medications will be allowed during the study).
6. Has an alanine aminotransferase (ALT) level <3*upper limit of normal (ULN) or an ALT level <5 *ULN with a confirmed diagnosis of nonalcoholic fatty liver disease (NAFLD).7. Does not plan to leave the geographic area within 1 calendar year following randomization.

For participants who have had the diagnosis of T2DM for less than 1 year and/or who are taking insulin prior to randomization, the following criteria must also be met:

8. Must have a fasting C-peptide concentration>=0.6 nanogram per milliliter (ng/mL) (>=0.20 nanomole per liter [nmol/L]) (drawn at least 1 week after treatment for ketosis or acidosis, if applicable).

9. No presence of autoantibodies as documented by glutamic acid decarboxylase [GAD] 65 and islet antigen [IA]-2 antibodies below the upper limit of the normal reference ranges at randomization.

10. Have a body mass index (BMI) greater than (>) 85th percentile, documented at randomization.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 152 (Actual)
Dates: Start 2016-10-14 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2022-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (67):
- United States (34):
  - Arkansas Children's Hospital Research Institute, Little Rock, Arkansas
  - Children's Hospital Los Angeles, Los Angeles, California
  - Sherif Khamis, Palmdale, California
  - Lucile Packard Children's Hospital at Stanford University, Palo Alto, California
  - Touro University California, Vallejo, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Children's National Health System, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Nemours Childrens Specialty Care - Jacksonville, Jacksonville, Florida
  - Baptist Diabetes Associates Research, Miami, Florida
  - University of South Florida/USF Health, Tampa, Florida
  - Endocrine Consultants Research, Columbus, Georgia
  - Endocrine Consultants Research - Oak Hill Court, Newnan, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kentucky Health Care, Lexington, Kentucky
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - University of Minnesota Masonic Children's Hospital - Pediatric Specialty Care Discovery Clinic, Minneapolis, Minnesota
  - Gulfside Clinical Research, Gulfport, Mississippi
  - Saint Louis University, St Louis, Missouri
  - Horizon View Medical Center, Las Vegas, Nevada
  - Saint Joseph's Regional Medical Center - Paterson, Paterson, New Jersey
  - University of Rochester, Rochester, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Greenville Health System - Patewood, Greenville, South Carolina
  - Monument Health Clinical Research, Rapid City, South Dakota
  - UT Le Bonheur Pediatric Specialists, Memphis, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine Advanced Liver Therapies, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Multicare Health System Institute for Research and Innovation, Tacoma, Washington
- Brazil (4):
  - Instituto de Estudos e Pesquisas Clinicas do Ceara, Fortaleza, Ceará
  - Hospital Universitario Joao de Barros Barreto, Belém, Pará
  - Instituto da Crianca com Diabetes, Porto Alegre, Rio Grande do Sul
  - Hospital Sirio Libanes, São Paulo
- Israel (3):
  - The Chaim Sheba Medical Center, Ramat Gan, Tel Aviv
  - Hadassah University Hospital Mount Scopus, Jerusalem
  - Clalit Medical Center, Tel Aviv
- Italy (4):
  - Ospedale Policlinico SS Annunziata, Chieti
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedaliero Universitaria Policlinico Paolo Giaccone, Palermo
  - Ospedale Pediatrico Bambino Gesu, Roma
- Mexico (11):
  - Endo Clinic, Guadalajara, Jalisco
  - Desarrollo Etico en Investigacion Clinica, Guadalajara, Jalisco
  - Investigacion Biomedica para el Desarrollo de Farmacos S.A. de C.V., Zapopan, Jalisco
  - Instituto Nacional de Pediatria, Mexico City, Mexico City
  - Mentrials, SA de CV, Mexico City, Mexico City
  - Centro de Atencion e Investigacion en Factores de Riesgo Cardiovascular Omega (Clinica Omega), Mexico City, Mexico City
  - IECSI-Centro Medico y de Investigacion Clinica, Monterrey, Nuevo León
  - Centro Integral Medico Sjr, San Juan del Río, Querétaro
  - Ono Consultoria Medica Integral, Aguascalientes
  - Centro de Investigacion Cardiometabolica de Aguascalientes, Aguascalientes
  - EL CIELO Medical Center, Puebla City
- Poland (5):
  - MedPolonia, Poznan, Greater Poland Voivodeship
  - Specjalistyczna Praktyka Lekarska ASPIRO, Wroclaw, Lower Silesian Voivodeship
  - Twoja Przychodnia - Centrum Medyczne Nowa Sol, Nowa Sól, Lubusz Voivodeship
  - Holmed, Warsaw, Masovian Voivodeship
  - Sonomed, Szczecin, West Pomeranian Voivodeship
- Russia (6):
  - Saint Petersburg State Pediatric Medical Academy, Saint Petersburg, Sankt-Peterburg
  - Republican Children's Clinical Hospital-Izhevsk, Izhevsk, Udmurtiya Republic
  - Kuzbass Regional Clinical Hospital n.a. S.V. Belyaev, Kemerovo
  - Novosibirsk State Medical University, Novosibirsk
  - Omsk Regional Children's Hospital, Omsk
  - Siberian State Medical University, Tomsk

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect Participant privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Peng XV, Klingensmith G, Hsia DS, Xie Y, Czerniak R, Tamborlane WV, Shah AS. A Randomized Phase 3 Study Evaluating the Efficacy and Safety of Alogliptin in Pediatric Participants with Type 2 Diabetes Mellitus. Diabetes Ther. 2025 May;16(5):865-883. doi: 10.1007/s13300-025-01700-3. Epub 2025 Mar 4. PMID 40032809

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 152 participants took part in the study at 67 investigative sites in Mexico, United States, Brazil, Israel, Italy and Russia from 14 October 2016 to 14 February 2022.
Pre-assignment Details: Participants with type 2 diabetes mellitus were enrolled to receive placebo or alogliptin 25 mg in a 1:1 ratio in this study.
Period: Overall Study
Arm/Group | Placebo | Alogliptin 25 mg
Started | 77 | 75
Safety Population (Safety Population included all participants who took at least 1 dose of study medication. One participant was randomized in error and did not receive any study medication.) | 76 | 75
Completed (Data is reported for participants who completed all study visits.) | 66 | 60
Not Completed | 11 | 15
Not completed — Pretreatment Event/Adverse Event | 1 | 0
Not completed — Significant Protocol Deviation | 1 | 0
Not completed — Lost to Follow-up | 3 | 5
Not completed — Voluntary Withdrawal | 3 | 5
Not completed — Pregnancy | 0 | 1
Not completed — Principal Investigator Discretion | 2 | 1
Not completed — Randomized but not Treated | 1 | 0
Not completed — Did not Complete Study but Contacted at Week 52 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Safety Set included all participants who took at least 1 dose of study medication.
Groups:
- Placebo: Alogliptin matching-placebo tablets, orally, QD for 52 weeks and background antidiabetic therapy (metformin and/or insulin), if applicable, maintained at the same dose throughout the first 26 weeks of the treatment period.
- Total: Total of all reporting groups
Arm/Group | Placebo | Alogliptin 25 mg | Total
Number analyzed (Participants) | 76 | 75 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.3 (2.21) | 14.2 (1.92) | 14.2 (2.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 53 | 104
  Male | 25 | 22 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 9 | 15
  Not Hispanic or Latino | 31 | 26 | 57
  Unknown or Not Reported | 39 | 40 | 79
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 14 | 11 | 25
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 16 | 32
  White | 44 | 44 | 88
  More than one race | 1 | 4 | 5
  Unknown or Not Reported | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: centimetres (cm)] | 164.7 (9.54) | 163.1 (8.79) | 163.9 (9.18)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 92.23 (26.826) | 90.72 (28.815) | 91.48 (27.749)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI was calculated as weight (kg) divided by square of height (m^2).
  kg/m^2 | 33.632 (7.8581) | 33.669 (8.6592) | 33.650 (8.2381)
Baseline of Glycosylated Hemoglobin (HbA1c) [Mean (Full Range); unit: percentage of HbA1c] — HbA1c is defined as the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound.
  percentage of HbA1c | 8.11 [5.7 to 11.3] | 8.16 [6.3 to 11.5] | 8.13 [5.7 to 11.5]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 26
Description: Change in the value of HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) was collected at Week 26 relative to Baseline. Mixed model for repeated measures (MMRM) was used for the analysis.
Time Frame: Baseline and Week 26
Population: FAS included all randomized participants in the safety set. Overall number of participants analyzed are the number of participants available for analysis.
Measure: Least Squares Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Placebo | Alogliptin 25 mg
Number analyzed (Participants) | 56 | 54
percentage of HbA1c | -0.011 (0.2809) | 0.091 (0.2879)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 25 mg; Test type: Superiority; p = 0.782, MMRM — P-values was assessed at 0.05 significance level using MMRM; Least Square (LS) Mean Difference = 0.102, 95% CI 2-sided [-0.627 to 0.831], Standard Deviation 0.3677 — MMRM:Treatment,scheduled visit,antidiabetic therapy,visit-by-treatment interaction-categorical effects;Baseline HbA1c,visit-by-baseline HbA1c interaction-continuous covariates;unstructured covariance matrix for correlation of repeated measurements

2. Secondary Outcome: Change From Baseline in HbA1c at Weeks 12, 18, 39 and 52
Description: Change in the value of HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) was collected at Weeks 12, 18, 39 and 52 relative to Baseline. MMRM was used for the analysis.
Time Frame: Baseline and Weeks 12, 18, 39 and 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Placebo | Alogliptin 25 mg
Number analyzed (Participants) | 62 | 62
percentage of HbA1c
  Change From Baseline at Week 12 | -0.319 (0.2173) | -0.365 (0.2223)
  Change From Baseline at Week 18: number analyzed (Participants) | 61 | 54
  Change From Baseline at Week 18 | -0.206 (0.2458) | -0.202 (0.2529)
  Change From Baseline at Week 39: number analyzed (Participants) | 47 | 49
  Change From Baseline at Week 39 | 0.502 (0.2802) | 0.091 (0.2866)
  Change From Baseline at Week 52: number analyzed (Participants) | 39 | 39
  Change From Baseline at Week 52 | 0.764 (0.3118) | 0.281 (0.3199)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 25 mg; Change From Baseline at Week 12; Test type: Superiority; p = 0.863, MMRM — P-values was assessed at 0.05 significance level using MMRM; LS Mean Difference = -0.046, 95% CI 2-sided [-0.567 to 0.476], Standard Deviation 0.2635 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg; Change From Baseline at Week 18; Test type: Superiority; p = 0.990, MMRM — P-values was assessed at 0.05 significance level using MMRM; LS Mean Difference = 0.004, 95% CI 2-sided [-0.614 to 0.622], Standard Deviation 0.3123 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Alogliptin 25 mg; Change From Baseline at Week 39; Test type: Superiority; p = 0.264, MMRM — P-values was assessed at 0.05 significance level using MMRM; LS Mean Difference = -0.412, 95% CI 2-sided [-1.139 to 0.316], Standard Deviation 0.3664 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Alogliptin 25 mg; Change From Baseline at Week 52; Test type: Superiority; p = 0.250, MMRM — P-values was assessed at 0.05 significance level using MMRM; LS Mean Difference = -0.483, 95% CI 2-sided [-1.314 to 0.348], Standard Deviation 0.4165 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants With Clinically Significant Physical Examination Findings
Description: Physical examination included examination of the following body systems: (1) respiratory system; (2) cardiovascular system; (3) nervous system (4) dermatologic system; and (5) gastrointestinal system. A summarized data for the above body systems was reported for participants with clinically significant findings.
Time Frame: From Day 1 to end of treatment period (up to 52 weeks)
Population: Safety Set included all participants who took at least 1 dose of study medication. Number analyzed is the number of participants available for analysis at the specific time point. Overall number of participants analyzed are the number of participants available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alogliptin 25 mg
Number analyzed (Participants) | 71 | 71
percentage of participants
  Week 4: number analyzed (Participants) | 1 | 0
  Week 4 | 0 |
  Week 12 | 0 | 0
  Week 18: number analyzed (Participants) | 2 | 1
  Week 18 | 0 | 0
  Week 26: number analyzed (Participants) | 69 | 68
  Week 26 | 0 | 0
  Week 32: number analyzed (Participants) | 3 | 0
  Week 32 | 0 |
  Week 39: number analyzed (Participants) | 66 | 67
  Week 39 | 0 | 0
  Week 45: number analyzed (Participants) | 2 | 0
  Week 45 | 0 |
  Week 52: number analyzed (Participants) | 57 | 50
  Week 52 | 0 | 0

4. Secondary Outcome: Percentage of Participants With Abnormal Vital Signs Values
Description: Vital signs included body temperature (oral or tympanic measurement), respiratory rate, blood pressure [systolic blood pressure (SBP) and diastolic blood pressure (DBP)] resting more than 5 minutes, and pulse (beats per minute). Data for participants with abnormal vital signs was reported. The percentage of participants are calculated based on the participants with non-missing data at that time-point.
Time Frame: From Day 1 to end of treatment period (up to 52 weeks)
Population: Safety Set included all participants who took at least 1 dose of study medication. Number analyzed are the number of participants with data available for analysis for given category. The percentages are rounded off to the next decimal value.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alogliptin 25 mg
Number analyzed (Participants) | 76 | 75
percentage of participants
  SBP (millimeters of mercury [mmHg]): >150: number analyzed (Participants) | 75 | 72
  SBP (millimeters of mercury [mmHg]): >150 | 1.3 | 2.8
  DBP (mmHg): >95: number analyzed (Participants) | 75 | 72
  DBP (mmHg): >95 | 4.0 | 4.2
  Pulse Rate (beats per minute [bpm]): <50: number analyzed (Participants) | 0 | 72
  Pulse Rate (beats per minute [bpm]): <50 |  | 1.4
  Pulse Rate (beats per minute [bpm]): >120: number analyzed (Participants) | 0 | 72
  Pulse Rate (beats per minute [bpm]): >120 |  | 1.4
  Temperature (Celsius [C]): <35.6: number analyzed (Participants) | 0 | 65
  Temperature (Celsius [C]): <35.6 |  | 3.1

5. Secondary Outcome: Percentage of Participants With Abnormal 12-lead Electrocardiogram (ECG) Findings
Time Frame: Week 26 and 52
Population: Safety Set included all participants who took at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | Alogliptin 25 mg
Number analyzed (Participants) | 76 | 75
participants
  Week 26: Abnormal, Not Clinically Significant | 7 | 6
  Week 26: Abnormal, Clinically Significant | 2 | 0
  Week 52: Abnormal, Not Clinically Significant | 7 | 6
  Week 52: Abnormal, Clinically Significant | 1 | 0

6. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAE)
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment.
Time Frame: From the study start up to end of the study (up to 54 weeks)
Population: Safety Set included all participants who took at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alogliptin 25 mg
Number analyzed (Participants) | 76 | 75
percentage of participants | 76.3 | 80.0

7. Secondary Outcome: Percentage of Participants With Total, Urinary and Respiratory Tract Infections and Hypersensitivity Reactions
Description: The percentage of participants are calculated based on the participants with non-missing data at that time-point.
Time Frame: From Day 1 to end of treatment period (up to 52 weeks)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alogliptin 25 mg
Number analyzed (Participants) | 76 | 75
percentage of participants
  Bladder Infection: number analyzed (Participants) | 76 | 9
  Bladder Infection | 0.0 | 11.1
  COVID-19 Infection: number analyzed (Participants) | 11 | 75
  COVID-19 Infection | 9.1 | 0.0
  Low Urinary Tract Infection: number analyzed (Participants) | 76 | 9
  Low Urinary Tract Infection | 0.0 | 11.1
  Lower Respiratory Tract Infection: number analyzed (Participants) | 11 | 9
  Lower Respiratory Tract Infection | 9.1 | 11.1
  Sinus Infection: number analyzed (Participants) | 11 | 9
  Sinus Infection | 9.1 | 11.1
  Upper Respiratory Infection: number analyzed (Participants) | 11 | 9
  Upper Respiratory Infection | 18.2 | 44.4
  Upper Respiratory Tract Infection: number analyzed (Participants) | 11 | 9
  Upper Respiratory Tract Infection | 9.1 | 0.0
  Lower Urinary Tract Infection: number analyzed (Participants) | 11 | 9
  Lower Urinary Tract Infection | 9.1 | 0.0

8. Secondary Outcome: Percentage of Participants With Hypoglycemia
Description: Mild to moderate hypoglycemia (abnormal low blood sugar) was defined as blood glucose less than (<) 60 milligram per deciliter (mg/dL) (3.33 millimole per liter [mmol/L]) in the presence of symptoms, or blood glucose <50 mg/dL (2.78 mmol/L) with or without symptoms. Severe hypoglycemia was defined as any episode requiring the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions, associated with a documented blood glucose <60 mg/dL (3.33 mmol/L) (unless the clinical situation makes obtaining a blood glucose difficult [example, it involves coma or seizure]).
Time Frame: From Day 1 to end of treatment period (up to 52 weeks)
Population: Safety Set included all participants who took at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alogliptin 25 mg
Number analyzed (Participants) | 76 | 75
percentage of participants | 7.9 | 5.3

9. Secondary Outcome: Percentage of Participants With Abnormal Safety Laboratory Findings
Description: The percentage of participants with any abnormal standard safety laboratory values (hematology, serum chemistry, and urinalysis) were collected throughout study. Abnormal values for hematology included hematocrit (percentage of hematocrit [%]), hemoglobin (grams per liter [g/L]), erythrocyte mean corpuscular volume (MCV)(femtoliter [fL]), erythrocytes (10^12/L), and leukocytes (10^9/L). Abnormal values for serum chemistry included for alanine aminotransferase (units per liter [U/L]), aspartate aminotransferase (U/L), cholesterol (millimoles per liter [mmol/L]), gamma glutamyl transferase (U/L), glucose (mmol/L): < 2.8 mmol/L, potassium (mmol/L), sodium (mmol/L), and triglycerides (mmol/L). ULN is upper limit of normal and LLN is lower limit of normal.
Time Frame: From Day 1 to end of treatment period (up to 52 weeks)
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alogliptin 25 mg
Number analyzed (Participants) | 75 | 73
percentage of participants
  Alanine Aminotransferase (U/L): >= 3 x ULN: number analyzed (Participants) | 75 | 72
  Alanine Aminotransferase (U/L): >= 3 x ULN | 10.7 | 5.6
  Aspartate Aminotransferase (U/L): >= 3 x ULN: number analyzed (Participants) | 75 | 0
  Aspartate Aminotransferase (U/L): >= 3 x ULN | 2.7 |
  Cholesterol (mmol/L): >7.72 mmol/L: number analyzed (Participants) | 75 | 72
  Cholesterol (mmol/L): >7.72 mmol/L | 1.3 | 1.4
  Gamma Glutamyl Transferase (U/L): >= 3 x ULN: number analyzed (Participants) | 75 | 72
  Gamma Glutamyl Transferase (U/L): >= 3 x ULN | 2.7 | 6.9
  Glucose (mmol/L): < 2.8 mmol/L | 13.3 | 20.5
  Glucose (mmol/L): >19.4 mmol/L | 10.7 | 13.7
  Potassium (mmol/L): <3.0 mmol/L: number analyzed (Participants) | 0 | 72
  Potassium (mmol/L): <3.0 mmol/L |  | 1.4
  Phosphate (mmol/L): >2.00 mmol/L: number analyzed (Participants) | 0 | 72
  Phosphate (mmol/L): >2.00 mmol/L |  | 1.4
  Sodium (mmol/L): <130 mmol/L: number analyzed (Participants) | 75 | 0
  Sodium (mmol/L): <130 mmol/L | 1.3 |
  Triglycerides (mmol/L): >2.5x ULN: number analyzed (Participants) | 75 | 72
  Triglycerides (mmol/L): >2.5x ULN | 6.7 | 1.4
  Hematocrit (%): >1.2 x ULN: number analyzed (Participants) | 74 | 72
  Hematocrit (%): >1.2 x ULN | 9.5 | 8.3
  Hemoglobin (g/L): < 0.8 x LLN: number analyzed (Participants) | 0 | 72
  Hemoglobin (g/L): < 0.8 x LLN |  | 1.4
  Hemoglobin (g/L): >1.2 x ULN: number analyzed (Participants) | 74 | 72
  Hemoglobin (g/L): >1.2 x ULN | 4.1 | 2.8
  Erythrocyte Mean Corpuscular Volume (fL): <70 fL: number analyzed (Participants) | 74 | 72
  Erythrocyte Mean Corpuscular Volume (fL): <70 fL | 2.7 | 2.8
  Erythrocyte Mean Corpuscular Volume (fL): >100 fL: number analyzed (Participants) | 0 | 72
  Erythrocyte Mean Corpuscular Volume (fL): >100 fL |  | 2.8
  Erythrocytes (10^12/L): >1.2 x ULN: number analyzed (Participants) | 74 | 72
  Erythrocytes (10^12/L): >1.2 x ULN | 1.4 | 1.4
  Leukocytes (10^9/L): >1.5 x ULN: number analyzed (Participants) | 74 | 72
  Leukocytes (10^9/L): >1.5 x ULN | 2.7 | 2.8

10. Secondary Outcome: Change From Baseline in Biomarkers of Bone Turnover at Weeks 26 and 52
Description: Biomarkers of bone turnover are bone-specific alkaline phosphatase to assess changes in bone formation and C-terminal telopeptide (CTX) to assess changes in bone resorption.
Time Frame: Baseline, Weeks 26 and 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Placebo | Alogliptin 25 mg
Number analyzed (Participants) | 67 | 68
units per liter (U/L)
  Baseline | 62.09 (37.084) | 62.62 (43.180)
  Change From Baseline at Week 26: number analyzed (Participants) | 60 | 59
  Change From Baseline at Week 26 | -6.20 (18.021) | -7.47 (20.139)
  Change From Baseline at Week 52: number analyzed (Participants) | 49 | 44
  Change From Baseline at Week 52 | -14.36 (18.000) | -15.43 (22.497)

11. Secondary Outcome: Change From Baseline in CD26 (CD4+T Cells) Surface Antigen Levels at Weeks 26 and 52
Time Frame: Baseline, Weeks 26 and 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of CD4+ T cells
Arm/Group | Placebo | Alogliptin 25 mg
Number analyzed (Participants) | 57 | 58
percentage of CD4+ T cells
  Baseline | 78.2 (8.60) | 77.7 (7.23)
  Change From Baseline at Week 26: number analyzed (Participants) | 45 | 42
  Change From Baseline at Week 26 | 1.2 (6.00) | 1.6 (7.20)
  Change From Baseline at Week 52: number analyzed (Participants) | 35 | 32
  Change From Baseline at Week 52 | 1.0 (5.39) | 0.8 (4.89)

12. Secondary Outcome: Change From Baseline in CD26 (CD8+T Cells) Surface Antigen Levels at Weeks 26 and 52
Time Frame: Baseline, Weeks 26 and 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of CD8+ T cells
Arm/Group | Placebo | Alogliptin 25 mg
Number analyzed (Participants) | 58 | 58
percentage of CD8+ T cells
  Baseline | 59.7 (13.51) | 59.6 (15.30)
  Change From Baseline at Week 26: number analyzed (Participants) | 46 | 41
  Change From Baseline at Week 26 | -0.2 (9.15) | 1.7 (8.76)
  Change From Baseline at Week 52: number analyzed (Participants) | 36 | 32
  Change From Baseline at Week 52 | 1.0 (7.63) | -0.3 (10.51)

ADVERSE EVENTS:
Time Frame: From the study start up to end of the study (up to 54 weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Safety Set included all participants who took at least 1 dose of study medication.
Arm/Group | Placebo | Alogliptin 25 mg
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/75
Serious Adverse Events (participants affected / at risk) | 3/76 | 2/75
Other Adverse Events (participants affected / at risk) | 39/76 | 31/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=76) | Alogliptin 25 mg (N=75)
Brain oedema (Nervous system disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1
Hypertensive urgency (Vascular disorders) | 1 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 1
Knee deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Lip injury (Injury, poisoning and procedural complications) | 1 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=76) | Alogliptin 25 mg (N=75)
Diarrhoea (Gastrointestinal disorders) | 7 | 7
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 5
Glycosylated haemoglobin increased (Investigations) | 4 | 0
Headache (Nervous system disorders) | 8 | 14
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 9
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 5 | 0
Influenza (Infections and infestations) | 0 | 7
Nausea (Gastrointestinal disorders) | 5 | 0
Sinusitis (Infections and infestations) | 4 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 5 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 4
Vomiting (Gastrointestinal disorders) | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.

DOCUMENTS (2):
  • Study Protocol (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT02856113/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT02856113/SAP_001.pdf